CLINICAL TRIAL: NCT01810237
Title: Validation of a Novel Dabigatran Based Peri-Operative Bridging Anticoagulation Protocol for Patients on Chronic Warfarin Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Sudeep Shivakumar, MD FRCPC, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SS001
Record Dates: First submitted 2013-02-28; First posted 2013-03-13 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thromboses
MeSH Terms: conditions — Venous Thrombosis | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dabigtran instead of LMWH for perioperative bridging. (Experimental)
  Interventions: Drug: Dabigatran.

INTERVENTIONS:
Drug: Dabigatran. — Dabigatran will be used instead of LMWH for anticoagulation bridging.

SUMMARY:
Research Questions:

1. Does using dabigatran bridging result in consistent therapeutic anticoagulation? What percentage of patients will become subtherapeutic on warfarin once dabigatran is stopped?
2. What is the incidence of bleeding events with the use of dabigatran overlapped with warfarin for bridging?
3. What is the cost benefit of using dabigatran instead of dalteparin for bridging anticoagulation?

DETAILED DESCRIPTION:
Subject Selection:

The study population will include low risk patients on long-term warfarin therapy for venous thromboembolic disease (VTE) followed by the hematology anticoagulation clinic. Low risk will be defined as status greater than 12 months post thromboembolic event.

The inclusion criteria include: (1) Low risk status as defined above, (2) Chronic warfarin therapy of at least 12 months duration with target INR of 2.0-3.0. Patients will be excluded from the study if one or more of the following are met: (1) increased risk of bleeding: bleeding requiring transfusion in last 12 months, history of hemorrhagic stroke or intracranial hemorrhage, recent gastrointestinal bleeding {<6 months}, history of a bleeding disorder, (2) Pregnant, breastfeeding or planning to become pregnant or breastfeed, (3) inhibitors allergy/sensitivity to dabigatran etexilate, (4)Creatinine Clearance < 30 mls/min, (5) Concomitant treatment with strong P-glycoprotein (6) Known thrombophilia including Factor V Leiden mutation, prothrombin gene mutation, antithrombin deficiency, protein C deficiency, protein S deficiency, and antiphospholipid antibody syndrome, and (7) inability to provide written informed consent.

Research Plan:

Patients will be identified by performing a manual search of the anticoagulation clinic database to identify patients on long-term warfarin therapy (>12 months). The results will be gleaned to identify patients who meet the inclusion criteria listed above.

Patients will then be contacted via phone by one of the anticoagulation clinic personnel who will be known to the patient and familiar with their history. If the patient is interested in participating in the study they will be asked to come in for an assessment to elucidate whether they meet inclusion criteria as described above. The coordinator will discuss the study principles, goals, and risks. If they are interested in the study informed consent will be obtained by the study coordinator, If they are not interested in participating in the study they will be excluded.

All patients enrolled in the study will undergo a planned sham surgery bridging protocol. This will take place for all patients over a 2 week period, which is the study period

On day -5, patients will stop taking their warfarin. They will have a baseline CBC, INR, activated partial thromboplastin time (aPTT), and thrombin time (TT) drawn. They will have an INR, aPTT and TT drawn daily for the duration of the study period, except the sham surgery day and the following day, until Day +5 post the sham surgery day or longer until the INR is = 2. If INR = 2 by Day -2 after stopping the warfarin, Vitamin K will be adminstered orally to help reversing the INR to normal. When the INR falls to <2.0, dabigatran will be started at a therapeutic dose of 150 mg orally twice daily. This will continue until the sham surgery day,. On the evening of the sham surgery day, warfarin will be restarted at twice the patient's maintenance dose to a maximum of 10 mg orally. Dabigatran will be decreased to a prophylactic dose of 150 mg orally daily. Warfarin dosing will be adjusted for each patient based on the day +2 INR. Dabigatran prophylaxis will continue until the INR is greater or equal to 2.0, at which point it will be discontinued and warfarin maintained. The INR will be checked the day after dabigatran is discontinued.

Basic demographic information will be collected from the study participants including age and sex. Patient's weight, medical history, current medications, and indication for long-term warfarin therapy will be recorded.

Safety Reporting The study will closely follow laboratory testing as it relates to coagulation status (INR, pTT, PTT, and CBC). All serious adverse events will be captured and appropriately assessed by the Principal Investigator as to causality and expectedness.

An adverse drug reaction is any noxious and unintended response to the study drug that is caused by administration of the drug. Lack of efficacy is not considered an adverse drug reaction. Untoward medical occurrences will be considered adverse drug reactions if a causal relationship between the event and the study drug cannot be ruled out.

An adverse event considered "serious" if it meets any of the following criteria:

* Results in death,
* Is life-threatening,
* Requires in-patient hospitalization or prolongation of existing hospitalization,
* Results in persistent or significant disability / incapacity,
* Is a congenital anomaly / birth defect, or
* Is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above.

Should any serious unexpected adverse drug reactions occur, it will be reported to Health Canada in accordance with the Regulations Amending the Food & Drug Regulations (1024 - Clinical Trials), Section C.05.014.

* Where it is neither fatal nor life-threatening, within 15 days after becoming aware of the information
* Where it is fatal or life-threatening, immediately where possible and, in any event, within 7 days after becoming aware of the information, and
* Within 8 days after having informed Health Canada of the ADR, submit as complete a report as possible which includes an assessment of the importance and implication of any findings.

All serious unexpected adverse drug reactions (and other safety events as applicable) will be reported to the Capital Health Research Ethics Board.

Analysis of data:

To address our primary objective, investigators will look at the percentage of patients in our cohort of 40 who have normal INR, on day 0 (sham surgery day) and thus would be ready to proceed with surgial intervention. Simple statistics will be used to calculate this percentage.

For patients who do not have corrected INR on day 0, and thus would have surgery delayed, a multivariate analysis to elucidate which factors contribute to insufficient normalization of bleeding tests will be performed.

Perioperative bridging anticoagulation with dabigatran and warfarin has not been studied previously, and investigators do not know the significance of the overlap on the INR. It is possible that patients will be under-anticoagulated in the post-operative period. An exploratory analysis will be performed to see if this is the case.

Lastly, a cost analysis will be performed comparing this dabigatran based bridging protocol with our current standard of care, a dalteparin based bridging protocol.

Confidentiality:

Patient information will be maintained in paper copy in the office of Dr. Sudeep Shivakumar in a locked cabinet. Only members of the study team will have access to this information. For the purposes of data-analysis, this information will be entered into a database within the CDHA firewall and will be password protected. Patients will be given a study identification number and therefore no identifiable information will be kept in the database. The study team will keep a list of screened and enrolled patients with corresponding study identification number. t

Once data analysis has been completed this information will be stored at the Capital Health Centre for Clinical Research in the Research Archive Room and then at an offsite storage facility leased by Capital Health (Iron Mountain, Hammonds Plains) for 25 years as per ICH-GCP Guidelines.

Drs. Shivakumar, McCurdy, Sharif, Anderson, and Shawwa are bound by physician-patient confidentiality.

Harms:

There is a theoretical risk of bleeding in this study, although exceedingly low.

There is a theoretical risk of bleeding when restarting warfarin while on prophylactic dabigatran. Bleeding laboratory parameters will be followed daily, except the day of Sham surgery and day 1, and this will allow us to detect any abnormalities in coagulation testing.

Lastly, there is a risk of allergy/sensitivity to Dabigatran.

Benefits:

There are three main benefits of this study:

1. Dabigatran offers an oral alternative to subcutaneous low molecular weight heparin. Subcutaneous injections can be painful and intimidating for many patients. An oral alternative is painless and easy to administer.
2. An increasing number of patients are being managed with dabigatran outside the context of clinical trials. No prior studies have evaluated dabigatran in the peri-operative setting and specifically the re-institution of warfarin.
3. LMWH regimens are very costly. Using the protocols as outlined above, the average cost per bridge in the LMWH regimen is $225.00 CDN whereas with Dabigatran it is $18.00 CDN, savings of $207.00 CDN per patient.

ELIGIBILITY:
Inclusion Criteria:

* Low risk status VTE
* Chronic warfarin therapy of at least 12 months duration with target INR of 2.0-3.0

Exclusion Criteria:

* Increased risk of bleeding: bleeding requiring transfusion in last 12 months, history of hemorrhagic stroke or intracranial hemorrhage, recent gastrointestinal bleeding {<6 months}, history of a bleeding disorder
* Pregnant, breastfeeding or planning to become pregnant or breastfeed
* Inhibitors allergy/sensitivity to dabigatran etexilate
* Creatinine Clearance < 30 mls/min
* Concomitant treatment with strong P-glycoprotein
* Known thrombophilia including Factor V Leiden mutation, prothrombin gene mutation, antithrombin deficiency, protein C deficiency, protein S deficiency, and antiphospholipid antibody syndrome
* Inability to provide written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Validation of a novel Dabigatran Based Peri-Operative Bridging Anticoagulation Protocol for Patients on Chronic Warfarin Therapy | 1 Year.